CLINICAL TRIAL: NCT03217188
Title: A Phase II Study of Proton Re-Irradiation for Recurrent Head and Neck Cancer
Brief Title: Proton Re-Irradiation for Recurrent Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-300
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Proton Re-Irradiation; 17-300
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a phase II study evaluating proton reirradiation for patients who have a recurrent or a second primary head and neck cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- fractionated full dose re-irradiation (Experimental)
  Interventions: Radiation: conventionally fractionated full dose re-irradiation
- hypofractionated palliative re-irradiation (Experimental)
  Interventions: Radiation: hypofractionated palliative re-irradiation

INTERVENTIONS:
Radiation: conventionally fractionated full dose re-irradiation — re-irradiation [60-70 Gy (RBE) in 2 Gy (RBE) fractions
  Arms: fractionated full dose re-irradiation
Radiation: hypofractionated palliative re-irradiation — course or a hypofractionated palliative re-irradiation "Quad Shot" course (3.7 Gy (RBE) twice daily x 2 days, followed by a 4 week break [+/- 2 weeks], repeated up to 4 cycles).
  Arms: hypofractionated palliative re-irradiation

SUMMARY:
The purpose of this study is to evaluate the tumor control and the side effects of using proton therapy for head and neck cancer that has come back.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to provide written informed consent
* Age ≥18 years at the time of consent
* Pathologically confirmed diagnosis of a recurrent or a new primary head and neck cancer
* A history of prior radiation to the head and neck (>/= 40 Gy, in 2 Gy/fraction equivalent)
* The recurrent or the second primary tumor is unresectable, the patient elects against surgical resection; patients who underwent surgery who has indications for postoperative radiation therapy is also eligible
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months after treatment Note: Patient with <6 months of life expectancy will be treated with palliative QUAD shot radiotherapy and those with > 6 months of life expectancy will be treated with conventionally fractionated full dose re-irradiation approach. Additional other factors determining which patients will be treated with Quad Shot therapy rather than full dose are if the patients have poor performance status, bulky or diffuse disease, significant medical co-morbidities, and significant metastatic disease burden.

Exclusion Criteria:

* Women who are pregnant or lactating
* Inability to comply with study and/or follow-up procedures
* <6 months between completion of prior RT and initiation of reirradiation using proton therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
locoregional recurrence-free | 12 months
  Locoregional recurrence includes events of local and/or regional recurrence, or death due to any cause. Patients who are lost to follow-up without any event may be removed from the protocol at the discretion of the principal investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm